CLINICAL TRIAL: NCT00564616
Title: A Randomized Controlled Study Focused on Impact of Adding Video Communication to Dispatch Instruction on the Quality of CPR, Including Chest Compressions and Rescue Breaths, in Simulated Cardiac Arrests
Brief Title: Simulation-Based Study of Adding Video Communication to Dispatch Instruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200708079R
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; video cell phone; dispatcher-assisted CPR
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- voice group (Placebo Comparator): the "voice group" received voice CPR instruction via a voice-only cell phone
  Interventions: Device: video cell phone
- video group (Experimental): the "video group" received interactive voice and video instruction via a video cell phone
  Interventions: Device: video cell phone

INTERVENTIONS:
Device: video cell phone — the "voice group" received voice CPR instruction via a voice-only cell phone, and the "video group" received interactive voice and video instruction via a video cell phone

SUMMARY:
The purpose of this study is to determine whether adding interactive video communication to dispatch instruction improves the quality of bystander cardiopulmonary resuscitation in simulated cardiac arrests.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) is a leading cause of adult death and bystander cardiopulmonary resuscitation (CPR) significantly improves survival. Dispatch assistance increases the chance of bystander CPR but the quality of dispatcher-assisted CPR (DA-CPR) remains unsatisfactory. This study is conducted to assess the effect of adding interactive video communication to dispatch instruction on the quality of bystander CPR, including chest compressions and rescue breathing, in simulated cardiac arrests.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers above 16 years of age who have not received any CPR training within the last 5 years were recruited.

Exclusion Criteria:

* Healthcare providers, non-Mandarin speaking individuals, and those with illness/physical conditions that prevent them from receiving telephone instructions or performing CPR were excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-04; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
quality of chest compressions and rescue breaths | every 30 seconds

SECONDARY OUTCOMES:
spent time to first effective chest compression and rescue breath | expressed as seconds

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Huei-Ming Ma, MD, PhD, Study Director — National Taiwan University Hospital

REFERENCES:
- [Background] Cheung S, Deakin CD, Hsu R, Petley GW, Clewlow F. A prospective manikin-based observational study of telephone-directed cardiopulmonary resuscitation. Resuscitation. 2007 Mar;72(3):425-35. doi: 10.1016/j.resuscitation.2006.07.025. Epub 2007 Jan 16. PMID 17224230
- [Derived] Yang CW, Wang HC, Chiang WC, Chang WT, Yen ZS, Chen SY, Ko PC, Ma MH, Chen SC, Chang SC, Lin FY. Impact of adding video communication to dispatch instructions on the quality of rescue breathing in simulated cardiac arrests--a randomized controlled study. Resuscitation. 2008 Sep;78(3):327-32. doi: 10.1016/j.resuscitation.2008.03.232. Epub 2008 Jun 25. PMID 18583016